CLINICAL TRIAL: NCT06579911
Title: Combining High-frequency Micro-ultrasound Target Biopsy and Multiparametric MRI Target Biopsy - Does It Increase the Detection Rate of Clinically Significant Prostate Cancer? a Prospective, Interventional, Single Centre, Randomized Controlled Trial
Brief Title: Combining High-frequency Micro-ultrasound and Multiparametric MRI Target Biopsy for Detecting Prostate Cancer
Acronym: Biopsy29
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Salzburger Landeskliniken (Other)
Responsible Party: Principal Investigator, Maximilian Pallauf, Biopsy29, Salzburger Landeskliniken
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Biopsy29
Record Dates: First submitted 2024-08-28; First posted 2024-08-30 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Prostatic Neoplasm of Uncertain Behavior
Keywords: Prostate cancer; prostate biopsy; high frequency ultrasound; fusion biopsy; multiparametric mri of prostate; pirads; primus
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants are randomly divided into two groups. One group (the experimental group) receives the combination of high-frequency micro-ultrasound, multiparametric MRI-targeted biopsy, and systematic biopsy. The other group (the control group) receives the current standard care, which includes only multiparametric MRI-targeted biopsy and systematic biopsy. This setup allows direct comparison of the detection rates of clinically significant prostate cancer between the new combination of interventions and the standard approach.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group U (Experimental): Use of high-frequency micro-ultrasound target biopsy, multiparametric MRI target biopsy and systematic biopsy for tumor detection
  Interventions: Device: High-frequency micro-ultrasound target biopsy
- Group S (Active Comparator): Use of multiparametric MRI target biopsy and systematic biopsy (current standard of care) for tumor detection
  Interventions: Device: conventional Multiparametric MRT target biopsy

INTERVENTIONS:
Device: High-frequency micro-ultrasound target biopsy — 1. High-frequency micro-ultrasound (transrectal ultrasound, 29 Hz, ExactVu) of the prostate. If suspicious lesions (PRIMUS >= 3) other than those already detected in multiparametric MRI are found, target biopsy will be performed. Maximum of four cores per lesion.
  2. Multiparametric MRI target biopsy (PI-RADS >= 3) of the prostate (transrectal ultrasound, 29 Hz, ExactVu). Maximum of four cores per lesion.
  3. Systematic biopsy (twelve cores) of the prostate
  Arms: Group U
Device: conventional Multiparametric MRT target biopsy — 1. Multiparametric MRT target biopsy (PI-RADS >= 3) of the prostate (conventional transrectal ultrasound, 8-10 Hz). Maximum of four cores per lesion.
  2. Systematic biopsy (twelve cores) of the prostate
  Arms: Group S

SUMMARY:
**Study Goal:** The purpose of this clinical trial is to determine if combining high-frequency micro-ultrasound with multiparametric MRI biopsy and a systematic biopsy can better detect clinically significant prostate cancer compared to current standard methods. This study is aimed at men who may have prostate cancer.

**Main Questions the Study Aims to Answer:**

1. Does the combination of new biopsy methods detect more clinically significant prostate cancers than the current standard method?
2. Does the new method not increase the detection of less serious forms of cancer beyond what the standard method detects?

**Participation in the Study:**

Participants in this study will undergo the following procedures:

* A high-frequency micro-ultrasound examination of the prostate.
* A multiparametric MRI-targeted biopsy of the prostate.
* A systematic biopsy of the prostate.

**Comparison Group:** Researchers will compare the new combination method with the current standard method to see if the new approach is more effective.

**Participants will:**

* Undergo several exams and biopsies depending on the results of previous tests.
* Attend regular follow-up appointments to monitor potential side effects and evaluate prostate health.
* Record their experiences and any symptoms in a diary.

DETAILED DESCRIPTION:
The primary objective of this study is (i) to demonstrate that the combination of highfrequency micro-ultrasound target biopsy, multiparametric MRI target biopsy, and systematic biopsy detects more clinically significant prostate cancer (>= ISUP 2) than multiparametric MRI target biopsy and systematic biopsy alone (current standard of care).

The secondary objective of this study is (ii) to demonstrate that the combination of high frequency micro-ultrasound target biopsy, multiparametric MRI target biopsy, and systematic biopsy does not detect more clinically insignificant prostate cancer (ISUP 1) than multiparametric MRI target biopsy and systematic biopsy alone (current standard of care).

The third objective of this study is (iii) to demonstrate that the combination of highfrequency micro-ultrasound target biopsy and multiparametric MRI target biopsy does not detect less clinically significant prostate cancer (>= ISUP 2) than multiparametric MRI target biopsy and systematic biopsy (current standard of care).

The fourth objective of this study is (iv) to demonstrate that the combination of highfrequency micro-ultrasound target biopsy and multiparametric MRI target biopsy detects less clinically insignificant prostate cancer (ISUP 1) than the combination of multiparametric MRI target biopsy and systematic biopsy (current standard of care).

ELIGIBILITY:
Inclusion Criteria:

- Men with suspected clinically significant prostate cancer, identified by the rise in PSA level, suspicious digital rectal examination or both and pathologic multiparametric MRI of the prostate (>= PI-RADS III)

Exclusion Criteria:

* Patients with histopathologic proven prostate cancer
* PSA > 20 ng/ml
* Finding in digital rectal examination >= cT2c
* Untreated bacterial infection of the prostate
* Untreated coagulopathy

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 400 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Detection of Clinically Significant Prostate Cancer via Prostate Biopsy | 2 Weeks
  This measure assesses whether participants have clinically significant prostate cancer (Gleason Score Sum ≥ ISUP 2) based on biopsy results, recorded as "yes" or "no".

SECONDARY OUTCOMES:
Detection of Clinically Insignificant Prostate Cancer via Prostate Biopsy | 2 Weeks
  This measure evaluates whether participants have clinically insignificant prostate cancer (Gleason Score Sum = ISUP 1) based on biopsy results, also recorded as "yes" or "no".

CONTACTS AND LOCATIONS:
Locations (1):
- Uniklinikum Salzburg, Department for Urology and Andrology, Salzburg, Salzburg, Austria

IPD SHARING:
Plan to Share IPD: No
No individual participant data (IPD) will be shared with other researchers. The data collected from participants will remain confidential and will be used exclusively for the analysis and reporting within the confines of this study. This approach ensures the privacy and security of participant information.

REFERENCES:
- [Background] Carioli G, Bertuccio P, Boffetta P, Levi F, La Vecchia C, Negri E, Malvezzi M. European cancer mortality predictions for the year 2020 with a focus on prostate cancer. Ann Oncol. 2020 May;31(5):650-658. doi: 10.1016/j.annonc.2020.02.009. Epub 2020 Apr 19. PMID 32321669
- [Background] Kim JK, Jang YJ, Cho G. Multidisciplinary functional MR imaging for prostate cancer. Korean J Radiol. 2009 Nov-Dec;10(6):535-51. doi: 10.3348/kjr.2009.10.6.535. PMID 19885309
- [Background] Kasivisvanathan V, Stabile A, Neves JB, Giganti F, Valerio M, Shanmugabavan Y, Clement KD, Sarkar D, Philippou Y, Thurtle D, Deeks J, Emberton M, Takwoingi Y, Moore CM. Magnetic Resonance Imaging-targeted Biopsy Versus Systematic Biopsy in the Detection of Prostate Cancer: A Systematic Review and Meta-analysis. Eur Urol. 2019 Sep;76(3):284-303. doi: 10.1016/j.eururo.2019.04.043. Epub 2019 May 24. PMID 31130434
- [Background] Rouviere O, Puech P, Renard-Penna R, Claudon M, Roy C, Mege-Lechevallier F, Decaussin-Petrucci M, Dubreuil-Chambardel M, Magaud L, Remontet L, Ruffion A, Colombel M, Crouzet S, Schott AM, Lemaitre L, Rabilloud M, Grenier N; MRI-FIRST Investigators. Use of prostate systematic and targeted biopsy on the basis of multiparametric MRI in biopsy-naive patients (MRI-FIRST): a prospective, multicentre, paired diagnostic study. Lancet Oncol. 2019 Jan;20(1):100-109. doi: 10.1016/S1470-2045(18)30569-2. Epub 2018 Nov 21. PMID 30470502
- [Background] Ghai S, Eure G, Fradet V, Hyndman ME, McGrath T, Wodlinger B, Pavlovich CP. Assessing Cancer Risk on Novel 29 MHz Micro-Ultrasound Images of the Prostate: Creation of the Micro-Ultrasound Protocol for Prostate Risk Identification. J Urol. 2016 Aug;196(2):562-9. doi: 10.1016/j.juro.2015.12.093. Epub 2016 Jan 12. PMID 26791931
- [Background] Rodriguez Socarras ME, Gomez Rivas J, Cuadros Rivera V, Reinoso Elbers J, Llanes Gonzalez L, Michel Mercado I, Fernandez Del Alamo J, Juarez Del Dago P, Sancha FG. Prostate Mapping for Cancer Diagnosis: The Madrid Protocol. Transperineal Prostate Biopsies Using Multiparametric Magnetic Resonance Imaging Fusion and Micro-Ultrasound Guided Biopsies. J Urol. 2020 Oct;204(4):726-733. doi: 10.1097/JU.0000000000001083. Epub 2020 Apr 21. PMID 32314932
- [Background] Abouassaly R, Klein EA, El-Shefai A, Stephenson A. Impact of using 29 MHz high-resolution micro-ultrasound in real-time targeting of transrectal prostate biopsies: initial experience. World J Urol. 2020 May;38(5):1201-1206. doi: 10.1007/s00345-019-02863-y. Epub 2019 Jul 15. PMID 31309290
- [Background] Laurence Klotz CM. Can high resolution micro-ultrasound replace MRI in the diagnosis of prostate cancer? Eur Urol Focus. 2020 Mar 15;6(2):419-423. doi: 10.1016/j.euf.2019.11.006. Epub 2019 Nov 24. PMID 31771935
- [Background] Cornud F, Lefevre A, Flam T, Dumonceau O, Galiano M, Soyer P, Camparo P, Barral M. MRI-directed high-frequency (29MhZ) TRUS-guided biopsies: initial results of a single-center study. Eur Radiol. 2020 Sep;30(9):4838-4846. doi: 10.1007/s00330-020-06882-x. Epub 2020 Apr 29. PMID 32350662
- [Background] Wiemer L, Hollenbach M, Heckmann R, Kittner B, Plage H, Reimann M, Asbach P, Friedersdorff F, Schlomm T, Hofbauer S, Cash H. Evolution of Targeted Prostate Biopsy by Adding Micro-Ultrasound to the Magnetic Resonance Imaging Pathway. Eur Urol Focus. 2021 Nov;7(6):1292-1299. doi: 10.1016/j.euf.2020.06.022. Epub 2020 Jul 9. PMID 32654967